CLINICAL TRIAL: NCT05300724
Title: A Multicenter, Prospective, Observational Study of the Progression of Intermediate Age-Related Macular Degeneration
Brief Title: An Observational Study of the Progression of Intermediate Age-Related Macular Degeneration
Acronym: HONU
Status: Active, not recruiting | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GE43220; 2022-000046-15 (EudraCT Number)
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intermediate AMD: Participants with iAMD will be evaluated for the progression of iAMD to more advanced atrophic AMD stages, such as nascent geographic atrophy (nGA) or incomplete retinal pigment epithelium and outer retinal atrophy (iRORA), and subsequently from nGA or iRORA to complete retinal pigment epithelium (cRORA) and outer retinal atrophy or geographic atrophy (GA), on Day 1 and thereafter every 12 weeks up to the end of the Observation Period, approximately 3 years.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered in this study.

SUMMARY:
This is a multicenter prospective study in participants with intermediate age-related macular degeneration (iAMD). One primary objective of this study is to assess iAMD disease progression, by the timeline and rates of conversion for high-risk iAMD at baseline to more advanced atrophic AMD stages. The other primary objective of this observational study is to assess the feasibility of measuring the rate of photoreceptor loss as a potential clinical endpoint. The study will consist of an observation period of approximately 3 years (~144 weeks) for participants.

ELIGIBILITY:
Inclusion Criteria:

* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, during the study for at least 28 days after the last fluorescein injection for the fluorescein angiography (FA) administration
* Study eye: High-risk intermediate AMD

Exclusion Criteria:

* Macular disease in either eye with subretinal deposits not typical of AMD
* Pigmentary abnormalities of the retina in either eye not typical of AMD
* Atrophy in either eye due to causes other than AMD
* Study eye: Any concurrent or history of ocular or intraocular condition
* Study eye: Intraocular surgery, including cataract surgery, within 3 months prior to Day 1
* Study eye: Retinal tears or peripheral retinal breaks within 3 months prior to Day 1
* Study eye: Concurrent or history of retinal laser photocoagulation or anti-vascular endothelial growth factor (anti-VEGF) treatment for exudative MNV, diabetic macular edema, retinal vein occlusion, or proliferative diabetic retinopathy
* Study eye: Presence of choroidal nevus with overlying drusen in the circle with a radius 3600 micrometer centered on the fovea
* Study eye: Previous participation in interventional clinical trials for GA or early stages of AMD, except for vitamins and minerals, regardless of the route of administration within the last 6 months, except for sham-arm participants
* Study eye: History of glaucoma surgery, corneal transplant, retinal pigment epithelium tear, retinal tear that involves the macula, retinal detachment
* Either eye: Uncontrolled progressive glaucoma
* Either eye: Moderate or severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy
* Either eye: History of recurrent infectious or inflammatory ocular disease
* Any concurrent or history of taking medications that can induce retinal toxicity

Ages: 50 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll participants with high risk intermediate AMD.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Conversion from iAMD to nGA /iRORA | Baseline up to 3 years
Rate of Conversion from nGA/iRORA to cRORA/GA | Baseline up to 3 years
Rate of Photoreceptor Loss as Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (74):
- United States (46):
  - Retina Partners of Northwest Arkansas, PLLC, Springdale, Arkansas
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants, San Diego, Poway, California
  - UC Davis Eye Center, Sacramento, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Southwest Retina Consultants, Durango, Colorado
  - Eye Care Center of Northern Colorado PC, Longmont, Colorado
  - Advanced Research, Coral Springs, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - New England Retina Consultants, Springfield, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Deep Blue Retina Clinical Research, Southaven, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Duke Eye Center, Durham, North Carolina
  - Cleveland Clinic Cole Eye Institute, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - EyeHealth Northwest, Portland, Oregon
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Tennessee Retina PC, Nashville, Tennessee
  - W Texas Retina Consultants PA, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Specialists, DeSoto, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (5):
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- France (5):
  - Centre Hospitalier Intercommunal, Créteil
  - Centre Ophtalmologique Pole Vision, Écully
  - CHU de GRENOBLE, Grenoble
  - Hôpital de La Croix Rousse, Lyon
  - Centre Ophtalmologique Maison-Rouge, Strasbourg
- Germany (8):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - University Medicine Gottingen Germany, Göttingen
  - Medizinische Hochschule Hannover, Innere Abteilung/Pneumologie, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinikum Munster, Münster
  - Augenzentrum am St Franziskus-Hospital, Münster
  - Universitatsklinikum Tubingen, Tübingen
- Israel (4):
  - Rambam Medical Center - PPDS, Haifa
  - Tel Aviv Sourasky Medical Center PPDS, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (5):
  - Azienda Sanitaria Universitaria Friuli Centrale ? PO Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Fondazione G.B. Bietti Per Lo Sudio E La Ricerca In Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Ospedale S. Giuseppe Multimedica, Milan, Lombardy
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan, Lombardy
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No